CLINICAL TRIAL: NCT04278612
Title: Evaluation of the Effectiveness of a Quality Improvement Intervention to Support Integration of Maternal, and Child and HIV Care in Primary Health Care Facilities in South Africa
Brief Title: Evaluation of the Effectiveness of a Quality Improvement Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: UNICEF (Other); Institute for Healthcare Improvement (Other)
Responsible Party: Principal Investigator, Christiane Horwood, Senior Researcher, University of KwaZulu
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: UNIP123
Record Dates: First submitted 2020-02-14; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Maternal and Child Health
Keywords: Quality improvement; Integrated care; Maternal health; Child health; HIV/AIDS; South Africa; Growth Monitoring; Child Growth; Nutrition
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The study evaluated 27 clinics in four sub-districts using a stepped-wedge design. Each sub-district received the intervention sequentially in a randomly selected order. Five waves of data collection were conducted in all participating clinics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Provision of comprehensive care including the following:
  Baby:
  Measure weight and length Plot on appropriate growth charts in Road to Health Card (RTHC) Discuss with mother about the growth of the baby Identification of malnutrition and appropriate management Age-appropriate nutrition counselling Immunisation Developmental screening Vitamin A supplementation Deworming HIV Care: If mother is HIV positive -
  * Polymerase chain reaction (PCR) test for the baby repeated at 10 weeks
  * Nevirapine for the baby for six weeks
  Mother:
  Cervical cancer screening Provide family planning Screening tuberculosis (TB) and sexually transmitted infections (STIs)
  HIV Care:
  * HIV positive mothers - provide ART for the mother and adherence support
  * HIV negative mothers- HIV test every three months while breastfeeding
  Interventions: Other: Quality improvement intervention to strengthen health service provision
- Control (Active Comparator): Routine maternal and child care service delivery
  Interventions: Other: Quality improvement intervention to strengthen health service provision

INTERVENTIONS:
Other: Quality improvement intervention to strengthen health service provision — Quality improvement intervention comprising of regular improvement meetings based at clinics.

SUMMARY:
This rigorous evaluation demonstrated that implementation of a time-limited quality improvement strategy effectively improved coverage of some components of an integrated maternal and child health service in a complex health environment, but we were unable to achieve the changes needed to provide a comprehensive package of care for mothers and children.

DETAILED DESCRIPTION:
Background: Despite policies and guidelines recommending integration of health services in South Africa, provision of maternal and child health services remains fragmented. This study evaluated a rapid, scaleable, quality improvement intervention to improve integration of maternal and child health and HIV services at a primary health level, in KwaZulu-Natal, South Africa.

Methods: A three-month intervention comprised of six quality improvement mentoring visits, learning sessions with clinic staff to share learnings, and a self-administered checklist aimed to assist health workers monitor and implement an integrated package of health services for mothers and children. The study evaluated 27 clinics in four sub-districts using a stepped-wedge design. Each sub-district received the intervention sequentially in a randomly selected order. Five waves of data collection were conducted in all participating clinics between December 2016-February 2017. A multi-level, mixed effects logistic regression was used to account for random cluster fixed time and group effects using Stata V13.1.

ELIGIBILITY:
Inclusion Criteria:

Women who attended the clinic for maternal and child health care services at 27 participating clinics from January 2016-February 2017.

Exclusion Criteria:

Women who did not attend the clinic for maternal and child health care services at 27 participating clinics from January 2016-February 2017.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women who attended the clinic for maternal and child health care services.
Enrollment: 1438 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2017-02-05 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Quality of Maternal and Child Care | 3 months
  Proportion of mother-baby pairs who received comprehensive care

SECONDARY OUTCOMES:
Quality of Child Care | 3 months
  Proportion of babies who receive growth monitoring services
Quality of Maternal Care | 3 months
  Proportion of mothers who receive feeding advice

IPD SHARING:
Plan to Share IPD: Yes
IPD will not be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Anytime
Access Criteria: We are more than happy to share our study protocol, statistical analysis plan or informed consent with anyone who is interested.

REFERENCES:
- [Derived] Haskins L, Chiliza J, Barker P, Connolly C, Phakathi S, Feeley A, Horwood C. Evaluation of the effectiveness of a quality improvement intervention to support integration of maternal, child and HIV care in primary health care facilities in South Africa. BMC Public Health. 2020 Mar 12;20(1):318. doi: 10.1186/s12889-020-8397-2. PMID 32164597